CLINICAL TRIAL: NCT01764269
Title: Assessing Fever Rates in Children Ages 24 to 59 Months After Live Attenuated Influenza Vaccine (LAIV) or Inactivated Influenza Vaccines (IIV) Using Text Messaging for U.S. Influenza Vaccines in 2012-2013 & 2013-2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAK8100
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inactivated influenza vaccine (IIV) (Other): Patients whose provider chooses to administer to them inactivated influenza vaccine (IIV)
  Interventions: Other: text message surveillance for fever
- Live attenuated influenza vaccine (LAIV) (Other): Patients whose provider chooses to administer to them Live attenuated influenza vaccine (LAIV)
  Interventions: Other: text message surveillance for fever

INTERVENTIONS:
Other: text message surveillance for fever

SUMMARY:
In this study, the investigators will prospectively assess fever rates in 24-59 month old patients during days 0-10 after administration of inactivated influenza vaccine (IIV) or live attenuated influenza vaccine (LAIV). Children in one of three study sites who receive these vaccines as part of their routine care can enroll in this study if their parent has the ability to receive and send text messages. Children enrolled in this study will be observed for an eleven day period starting on the day of vaccine administration via a series text messages to their parents.

ELIGIBILITY:
Inclusion Criteria:

1. are 24 through 59 months of age,
2. have a visit at a study site anytime during the study period,
3. receive first dose LAIV or IIV in the season,
4. the parent has a cell phone with text messaging capabilities, and
5. the parent speaks English or Spanish.

Exclusion criteria:

1. any chronic medical condition in the child that precludes receipt of LAIV (except for history of asthma or a wheezing episode within the past 12 months noted in the medical record),
2. currently on oral or other systemic steroids or used in the past month,
3. currently on inhaled steroids or used in the past 2 weeks,
4. presence of fever >=100.4 at time of vaccination,
5. administration of any antipyretic in the 6-hour period prior to vaccination,
6. stated intent, at time of vaccination, to use prophylactic antipyretics before the development of a fever,
7. parent only speaks a language other than English or Spanish,
8. parent's inability to read text messages,
9. child receiving the second dose of influenza vaccine in the current season.

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 656 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
fever | 11 days
  day of vaccination plus 10 more days

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Philip LaRussa, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Columbia University, New York, New York